CLINICAL TRIAL: NCT02411175
Title: The Efficacy of Individualised Homeopathic Treatment on Constipation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Johannesburg (Other)
Responsible Party: Principal Investigator, Dr J. Pellow, Dr J. Pellow, University of Johannesburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FarhanaNakhooda201007840
Record Dates: First submitted 2015-04-03; First posted 2015-04-08 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Constipation
Keywords: Constipation; Homeopathy
MeSH Terms: conditions — Constipation | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 20% Ethanol (Experimental): 20% ethanol will be medicated with the individualised homeopathic remedy as determined by the researcher and administered as drops. The potency, dose and frequency of the medicated 20% ethanol drops will be determined for each prescription, in accordance with the laws that govern homeopathic prescribing.
  Interventions: Other: Individualised Homeopathic Remedy; Drug: 20% ethanol

INTERVENTIONS:
Other: Individualised Homeopathic Remedy — 20% ethanol will be medicated with the Individualised Homeopathic Remedy in the potency determined by the researcher in accordance with the laws that govern individualised homeopathic prescribing. The medicated 20% ethanol will be administered as drops.
  Other Names: Similimum
Drug: 20% ethanol

SUMMARY:
Constipation is an umbrella term encompassing either infrequent bowel movements, difficult evacuation of stool, hard stool or a sensation of incomplete defecation. It affects 10-15% of the global population. Constipation may negatively impact physical health, moods and social life. There exists a 50% dissatisfaction with traditional approach of laxative use. Conventional laxatives only offer a temporary solution and may cause dependency. Side-effects of conventional laxatives include nausea, vomiting, flatulence, diarrhoea, abdominal pain, electrolyte imbalance and skin eruptions. Homeopathy is a potential treatment option for constipation, however further research is needed in this regard.

The aim of this study is to determine the efficacy of individualised homeopathic treatment on constipation using case studies, an adapted Bowel Function Diary and the Bristol Stool Form Scale.

DETAILED DESCRIPTION:
The research study will be of an embedded mixed method case study design and take place over a 6 week period at the University of Johannesburg Doornfontein Health Centre. Ten participants of either gender, between the ages of 18 to 50 years will be recruited using advertisements placed at the Doornfontein campus Health Centre.Those interested in participating in the research will be requested to attend an initial meeting in which they will receive a Participant Information Form and be requested to sign a Consent Form.

Participants meeting the inclusion criteria will be recruited into the study and a Selection Questionnaire confirming their constipation status will be completed with the help of the researcher. The researcher will then perform a full case taking and relevant physical examination of the participant, the details of which will be recorded on a homeopathic Case Taking Form, as designed by the researcher. The characteristic details of the case will then be identified and analysed using using the Mercurius software Repertory. The homeopathic Materia Medica will be referred to in order to confirm the remedy which best suits the presenting symptomology of the participant. The repertorisation and remedy selection will be conducted under the supervision of a qualified homeopath.

The potency, dose and frequency of the selected remedy will be determined according to the laws that govern individualised homeopathic prescribing.

The remedy will be administered along with an explanation and demonstration on how to take the remedy. A set of written instructions will be provided for the participant in the form of a Patient Information Leaflet.

The participant will be requested to monitor each defecation session and a Bowel Function Diary will be used to record the frequency of defecation, the stool form and the level of difficulty on passing a stool. Participants will return for three follow up consultations at 2 week intervals. If dramatic changes occur in the participant, they will be requested to contact the researcher, who will adjust the treatment accordingly.

At each follow up consultation, the participant's case will be re-evaluated with special attention made to changes in symptoms or the appearance of new symptoms, the details of which will be recorded on the Case Follow Up Form, as designed by the researcher. A remedy will be prescribed in the same manner as the initial consultation. The prescription may be repeated or altered in accordance with the participant's presenting symptoms and response to the previous prescription. The laws that govern individualised homeopathic prescribing will be used at all times in determining a prescription.

The qualitative data collected from the case taking forms, will be used by the researcher to write detailed case studies. The quantitative data collected, using the Bowel Function Diary and Bristol Stool Form Scale, will be used to assess the participants' changes in defecation quality and frequency over the course of treatment, the results of which will be represented graphically.

This study will contribute to the body of knowledge of the homeopathic treatment of constipation and may provide a foundation for further research on the efficacy of individualised homeopathic treatment of constipation.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 18-50 years,
* meet the Rome II criteria for constipation which lists:
* have a bowel evacuation for 3 or less times in a week, for the last 3 months OR
* have to strain, have hardened stool, or have incomplete bowel evacuation for at least 25% of the time, for the last 3 months.

Exclusion Criteria:

* People currently on treatment for their constipation,
* who have used laxatives more than three times in the past month,
* are on medications which have constipation as a side effect,
* with pre-diagnosed colon cancer, irritable bowel syndrome- constipation dominant, spastic colon or diverticulitis, and those who had a stroke, and,
* pregnant females.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Bowel Function Diary (Adapted) | 6 Weeks
  The Bowel Function Diary is a is a daily record of factors relating to defecation. For this study only two of its items will be monitored- the number of bowel movements and the associated ease or difficulty of defecation. The diary has been demonstrated to have an acceptable test-retest reliability and supported validity for each item, with a p-value of <0.001.

SECONDARY OUTCOMES:
Bristol Stool Form Scale | 6 Weeks
  The Bristol Stool Form Scale is a 7 score visual scale to measure stool consistency. It has been proved to be a reliable and valid measure, and can be effectively used with participants over the age of 8 for research purposes.
Means of case notes, recorded on homeopathic Case Taking Form | Every 2 weeks for 6 weeks
  Qualitative data will be collected by means of case notes, recorded on homeopathic Case Taking Forms, which will be taken at weeks 0, 2, 4 and 6.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Solomon, D.TechHom, Study Director — University of Johannesburg
Locations (1):
- University of Johannesburg, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No